CLINICAL TRIAL: NCT04001244
Title: Translational Research in Pelvic Pain. Deep Phenotyping of Women With Endometriosis-associated Pain and Bladder Pain Syndrome
Brief Title: Translational Research in Pelvic Pain
Acronym: TRiPP
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Boston Children's Hospital (Other); Michigan State University (Other); Bayer (Industry); Grünenthal GmbH (Industry); Esteve (Other); Queen Mary University of London (Other); Aalborg University (Other); Endometriosis.org (Unknown); International Painful Bladder Foundation (Unknown); Pelvic Pain Support Network (Unknown); King's College London (Other); Heidelberg University (Other); University of Edinburgh (Other); University of Jena (Other); Universität Münster (Other); Universidade do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: TRiPP WP9
Record Dates: First submitted 2019-05-16; First posted 2019-06-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis; Bladder Pain Syndrome; Chronic Pain
MeSH Terms: conditions — Endometriosis; Cystitis, Interstitial; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva Blood Urine Bladder biopsies (for BPS patients) Eutopic and ectopic endometrium (for endometriosis patients and Oxford controls)
  N.B. Biospecimens have already been collected for all Endometriosis (with and without bladder symptoms) and Control subjects, therefore new bio specimens are only being collected for the BPS cohort or if necessary for additional analyses (e.g. salivary cortisol), in which case samples will not be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Endometriosis (EAP): Surgical diagnosis of endometriosis (aim equal distribution of stage I/II and stage III/IV disease); at least one pelvic pain >3/10; pain not perceived by the patient as arising from the bladder; no urinary symptoms (e.g. urge, frequency)
- Bladder Pain Syndrome (BPS): Bladder pain syndrome (as defined by ESSIC criteria: pelvic pain, pressure or discomfort for greater than 6 months, perceived to be related to the urinary bladder accompanied by at least one other urinary symptom like persistent urge to void or frequency); no history of endometriosis
- Endometriosis and Bladder Pain (EABP): Surgical diagnosis of endometriosis; at least one pelvic pain >3/10; pain perceived by the patient as arising from the bladder AND from other area(s) of the pelvis; at least one urinary symptom (e.g. urge, frequency)
- Controls: No endometriosis; No pelvic pain (or dysmenorrhea; NRS <3/10)
- Pelvic Pain (PP): At least one pelvic pain >3/10; no endometriosis; pain not perceived by the patient as arising from the bladder; no urinary symptoms (e.g. urge, frequency)

SUMMARY:
This study aims to better understand the pathways leading to pain in women with two types of pelvic pain condition (endometriosis-associated pain and bladder pain syndrome) and determine whether these pathways can be used to subgroup patients.

DETAILED DESCRIPTION:
Chronic pelvic pain is as common as asthma, migraine and back pain and has a very significant impact on quality of life. However, it is still poorly understood and the available treatments are limited and often not successful. This project focuses on two causes of chronic pelvic pain: endometriosis and interstitial cystitis/bladder pain syndrome. Endometriosis (the presence of tissue resembling the lining of the womb outside of the womb) is very common, affecting ~1 in 10 women, and is associated with often disabling pelvic pain symptoms including painful periods, pain throughout the month, and pain associated with sex, passing urine and opening bowels. Interstitial cystitis/bladder pain syndrome is much less common but dramatically reduces quality of life with many women planning their day around trips to the toilet.

This multi-centre study will be carried out at 3 sites in Europe and 1 in the U.S.. Rather than focusing on the pelvis, the investigators will approach these conditions in the context of other chronic pain conditions with which they share many features and thus consider the many different systems that might contribute to generating and maintaining pain. The investigators will combine detailed clinical and questionnaire data with tests of the function of a variety of systems (including nerve function, stress response and psychology) and the results of analyses of different body fluids and tissues (including blood, urine, endometriosis lesions). No study treatment or intervention will be given during TRiPP. The aim is to identify pathways responsible for pain in these women and determine whether they can be divided into subgroups on the basis of different pain pathways that might therefore respond to different treatments. Ultimately the investigators hope to identify new targets for treatment and contribute to the design of more personalised treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 - 50 years.
* Participant is willing and able to give informed consent for participation in the study.
* EAP/EABP/CON: previously enrolled in EndOX or BCE cohorts with consent to be contacted again.
* EAP: Surgical diagnosis of endometriosis; at least one pelvic pain >3/10.
* EABP: Surgical diagnosis of endometriosis; at least one pelvic pain >3/10; pain perceived by the patient as arising from the bladder AND from other area(s) of the pelvis; at least one urinary symptom (e.g. urge, frequency).
* BPS: fulfil ESSIC criteria (Pelvic pain, pressure or discomfort for greater than 6 months, perceived to be related to the urinary bladder accompanied by at least one other urinary symptom like persistent urge to void or frequency).

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* EAP: pain perceived by the patient as arising from the bladder; urinary symptoms (e.g. urge, frequency).
* CON: previous diagnosis of endometriosis; pelvic pain or dysmenorrhoea (NRS>3/10)
* BPS: previous diagnosis of endometriosis.

Additionally, for physiological testing:

Exclusion:

• Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

And for fMRI:

Inclusion:

• fMRI compatible.

Exclusion:

* Contraindication to fMRI scan i.e. metallic implants, stents, clips, weight greater than acceptable for local fMRI scanner etc.
* Use of centrally acting drugs in the previous 3 months (e.g. anti-epileptics, anti-depressants, anxiolytics, gabapentin, pregabalin, duloxetine). N.B. Regular use of standard analgesics including opiates is not an exclusion criterion, however, women will be asked to refrain from taking such drugs for 8 hours prior to their brain scan if at all possible.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Controls, EAP and EABP will be selected from already recruited cohorts, with permission to be recontacted, in the ENDOX (University of Oxford) and BCE (Boston Childrens Hospital) studies. BPS will be recruited from secondary/tertiary care clinics and from adverts on patient support group sites and in local media.
Sampling Method: Non-Probability Sample
Enrollment: 787 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | 1 year
  QST of the dorsal of the foot and midline lower abdomen according to the German Neuropathic Pain Network Protocol.
Presence of abdominal wall muscle tenderness | 1 year
  Assessment of the abdominal wall specifically looking for muscle tenderness according to a standardised protocol (an enhanced Carnetts test as described by Scheltinga and Roumen 2017). Subjects will be categorised into muscle tenderness present or absent.
Change of pressure pain threshold (PPT) | 1 year
  A standardised conditioned pain modulation (CPM) paradigm will be used to investigate the change in pressure pain threshold on the dorsum of the foot. An ischaemic stimulus to the contralateral arm will be used as the conditioned stimulus. The foot PPT will be measured before the conditioned stimulus and immediately after. The change will be reported as the (PPTbefore - PPTafter).
Area under the curve (AUC) of single day salivary cortisol profile | 1 year
  Saliva will be collected at home at the specified times allowing a daily AUC of salivary cortisol for each subject to be calculated. Collection times: waking; 30-45 minutes after waking; before lunch; before dinner; bedtime.
Change in salivary cortisol | Saliva collected immediately before and immediately after CPM paradigm (outcome 3).
  A saliva sample will be collected at rest immediately before the CPM paradigm described in outcome 3 and then again immediately after. The ischaemic pain stimulus used as the conditioning stimulus in this paradigm is the most noxious component of the physiological testing paradigms used in this study and therefore the most likely to generate a stress response. The change will be reported as Cortisol(before)-Cortisol(after).
Heart rate (HR) | 1 year
  Assessed over a 20 minute period at rest.
Change in heart rate | HR assessed immediately before and immediately after the CPM paradigm (outcome 3)
  Assessed at rest immediately before the CPM paradigm described in outcome 3 and then again immediately after. The ischaemic pain stimulus used as the conditioning stimulus in this paradigm is the most noxious component of the physiological testing paradigms used in this study and therefore the most likely to generate a stress response. The change will be reported as HR(before) - HR(after).
Blood pressure (BP) | 1 year
  Assessed over a 20 minute period at rest. Measured in mmHG.
Change in Blood pressure | BP assessed immediately before and immediately after the CPM paradigm (outcome 3)
  Assessed at rest immediately before the CPM paradigm described in outcome 3 and then again immediately after. The ischaemic pain stimulus used as the conditioning stimulus in this paradigm is the most noxious component of the physiological testing paradigms used in this study and therefore the most likely to generate a stress response. The change will be reported as BP(before) - BP(after).
Bladder sensitivity to filling | 1 year
  Assessed with standardised non-invasive bladder filling paradigm, measured as time to verbal reports of different sensations of bladder fullness (first sensation, first urge) and then need to void (maximum tolerance) after drinking 600 ml water. Subjects will be categorised into those with bladder sensitivity compared to published norms for reproductive age women and those with normal bladder sensation.
Volume voided at maximum tolerance | 1 year
  Assessed with standardised non-invasive bladder filling paradigm described in outcome 10. The volume of urine voided when maximum tolerance is reached will be measured in mls.
fMRI scan | 1 year
  fMRI scan with response to punctate stimuli of midline lower abdomen.
Pain Catastrophising: Pain Catastrophising Scale (PCS) (Sullivan) | Baseline
  Measured with the Pain Catastrophising Scale (Sullivan). Scores range from 0 - 52 with high scores representing higher levels of pain catastrophising. Although three sub scales exist they will not be assessed for the purposes of these main analyses.
Comorbid psychological distress | Baseline
  Measured with the Hospital Anxiety and Depression Scale (HADS). Scores range from 0 - 21 for each of the two sub scales measuring anxiety and depression. The two sub scales will be summed as a unidimensional measure of psychological distress in initial analyses (0 - 42 with higher scores representing greater distress).

SECONDARY OUTCOMES:
Metabolomic data | Baseline
  Discovery study of levels of all known metabolite in plasma using an established validated proprietary tool designed by Metabolon (https://www.metabolon.com).
Proteomic data | Baseline
  Study measuring levels of proteins detected on two panels (inflammation and neurological) as designed by OLink (https://www.olink.com).
Transcriptomic data | Baseline
  Discovery transcriptomic analysis of matched eutopic and ectopic endometrium from endometriosis and control women will be performed on a subgroup of participants. Both descriptive data and pathway analysis will be performed.
Comorbidities | Baseline
  Assessed with the complex medical symptoms inventory (CMSI).
  The CMSI contains a 41 item symptom screener, which an increasing score on adds up to a higher functional somatic burden (scores range from 0-41). Additionally, clusters of symptoms point to specific diagnoses for which the full diagnostic criteria questions are provided allowing the commonest overlapping pain conditions to be screened for:
  Fibromyalgia temporomandibular disorders irritable bowel syndrome chronic tension type headache migraine chronic low back pain myalgic encephalitis/chronic fatigue syndrome interstitial cystitis/painful bladder syndrome endometriosis vulvodynia
Past trauma | Baseline
  Assessed with the Childhood Traumatic Events Scale (CTES). Scores range from 0 - 42 with higher scores representing more experience of early trauma. No sub scales will be derived.
Recent trauma | Baseline
  Assessed with the Recent Traumatic Events Scale (RTES). Scores range from 0 - 42 with higher scores representing more experience of recent trauma. No sub scales will be derived.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Vincent, DPhil, Principal Investigator — University of Oxford
Locations (2):
- IBMC, Porto, Portugal
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the study and all follow up analyses are complete de-identified data will be deposited in a publically accessible repository as required by the funders.
Supporting Information: Study Protocol
Time Frame: Data will be available once all analyses are complete.
Access Criteria: Data will be publically accessible

REFERENCES:
- See also: Project website as part of the overall project IMI-PainCare that TRiPP sits within — https://www.imi-paincare.eu/PROJECT/TRIPP/